CLINICAL TRIAL: NCT05339334
Title: A Phase 1, Single Center, Open-label Study of PF-07321332 Administrated as Multiple Oral Doses in Healthy Chinese Participants.
Brief Title: A Study to Learn About the Study Medicine PF-07321332 and Ritonavir in Adult Healthy Chinese Participants.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: C4671016
Record Dates: First submitted 2022-04-14; First posted 2022-04-21 (Actual); Results first posted 2024-10-08 (Actual); Last update posted 2024-10-08 (Actual); Status verified 2024-09

CONDITIONS: Healthy Participants
Keywords: severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2); coronavirus disease 2019 (COVID-19)
MeSH Terms: conditions — COVID-19 | interventions — nirmatrelvir and ritonavir drug combination

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- PF-07321332/ritonavir (Experimental): PF-07321332/ritonavir will be given by mouth two times a day for 10 days to adult Chinese healthy volunteers
  Interventions: Drug: PF-07321332/ritonavir

INTERVENTIONS:
Drug: PF-07321332/ritonavir — PF-07321332/ritonavir will be given by mouth two times a day for 10 days

SUMMARY:
The purpose of this Phase 1 clinical trial is to help us understand how the drug is changed and eliminated from your body after you take it, the safety, and the the extent to which dise effects can be tolerated of PF-07321332 when PF-07321332 and ritonavir are given to healthy adult Chinese participants.

ELIGIBILITY:
Inclusion Criteria:

* Healthy Chinese participants
* No clinical relevant abnormalities
* Body mass index (BMI):17.5-28

Exclusion Criteria:

* Any clinical significant illness
* History of alcohol abuse
* Use of prescription or nonprescription drugs and dietary and herbal supplements within 7 days prior the first study dose
* Abnormal clinical lab tests: aspartate aminotransferase (AST), alanine aminotransferase (ALT), total bilirubin, estimated glomerular filtration rate (eGFR)
* Abnormal vital signs, such 12-electrocardiogram (ECG), blood pressure and pulse rate
* Blood donation within 60 days
* History of human immunodeficiency virus (HIV), hepatitis B surface antigen (HBsAg), hepatitis B core antibody (HBcAb), hepatitis C antibody (HCVAb)
* Other medical or psychiatric may inappropriate for the study

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 14 (Actual)
Dates: Start 2022-03-10 (Actual); Primary Completion 2022-04-21 (Actual); Study Completion 2022-04-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Huashan Hospital,Fudan University, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=C4671016

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The study consisted of 1 treatment group: multiple oral doses of PF-07321332300 mg/ritonavir 100 mg. A total of 14 healthy participants were enrolled and treated.
Groups:
- PF-07321332 300 mg + Ritonavir 100 mg: The study interventions used in the study were PF-07321332 300 mg and ritonavir 100 mg, administered orally once every 12 hours (q12h) for a total of 19 doses (Day 1 to Day 10), with the last dose administered on the morning of Day 10 (no evening dose on Day 10).
Period: Overall Study
Arm/Group | PF-07321332 300 mg + Ritonavir 100 mg
Started | 14
Completed | 14
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: All participants who were enrolled in the study.
Arm/Group | PF-07321332 300 mg + Ritonavir 100 mg
Number analyzed (Participants) | 14
Age, Continuous [Mean (Standard Deviation); unit: years] | 33.1 (6.78)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 8
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 14
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 14
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 0
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: PF-07321332 Maximum Observed Plasma Concentration (Cmax) on Day 1
Description: Cmax is maximum plasma concentration .
Time Frame: Day 1 (pre-dose, 0.5, 1, 1.5, 2, 4, 6, 8, and 12 hours)
Population: The pharmacokinetic (PK) parameter analysis set was defined as all participants assigned to investigational product and treated who had at least 1 of the PK parameters of primary interest measured.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanograms per milliliter (ng/mL)
Arm/Group | PF-07321332 300 mg + Ritonavir 100 mg
Number analyzed (Participants) | 14
nanograms per milliliter (ng/mL) | 3082 (29)

2. Primary Outcome: PF-07321332 Maximum Observed Plasma Concentration (Cmax) on Day 10
Description: Cmax is maximum plasma concentration
Time Frame: Day 10 (pre-dose, 0.5, 1, 1.5, 2, 4, 6, 8 and 12 hours)
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanograms per milliliter (ng/mL)
Arm/Group | PF-07321332 300 mg + Ritonavir 100 mg
Number analyzed (Participants) | 14
nanograms per milliliter (ng/mL) | 4500 (14)

3. Primary Outcome: PF-07321332 Time for Maximum Observed Plasma Concentration (Tmax) on Day 1
Description: Tmax is the time for maximum plasma concentration
Time Frame: Day 1 (pre-dose, 0.5, 1, 1.5, 2, 4, 6, 8, and 12 hours)
Population: as for outcome 1
Measure: Median (Full Range); unit: hours (hr)
Arm/Group | PF-07321332 300 mg + Ritonavir 100 mg
Number analyzed (Participants) | 14
hours (hr) | 1.76 [1.00 to 4.00]

4. Primary Outcome: PF-07321332 Time for Maximum Observed Plasma Concentration (Tmax) on Day 10
Description: Tmax is the time for maximum plasma concentration
Time Frame: Day 10 (pre-dose, 0.5, 1, 1.5, 2, 4, 6, 8 and 12 hours)
Population: as for outcome 1
Measure: Median (Full Range); unit: hours (hr)
Arm/Group | PF-07321332 300 mg + Ritonavir 100 mg
Number analyzed (Participants) | 14
hours (hr) | 2.00 [1.00 to 4.02]

5. Primary Outcome: PF-07321332 Area Under the Plasma Concentration-time Profile From Time Zero to Time Point on 12 Hours (AUC12) on Day 1
Description: Area under the plasma concentration-time profile from time Zero to time point on 12 hours
Time Frame: Day 1 (pre-dose, 0.5, 1, 1.5, 2, 4, 6, 8, and 12 hours)
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram*hour per milliliter (ng*hr/mL)
Arm/Group | PF-07321332 300 mg + Ritonavir 100 mg
Number analyzed (Participants) | 14
nanogram*hour per milliliter (ng*hr/mL) | 19660 (26)

6. Primary Outcome: PF-07321332 Area Under the Plasma Concentration-time Profile From Time Zero to Time Tau (Where Tau=12 Hours) (AUCtau) on Day 10
Description: Area under the plasma concentration-time profile from time 0 to the time of the end of the dosing interval (tau), where tau=12 hours.
Time Frame: Day 10 (pre-dose, 0.5, 1, 1.5, 2, 4, 6, 8 and 12 hours)
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram*hour per milliliter (ng*hr/mL)
Arm/Group | PF-07321332 300 mg + Ritonavir 100 mg
Number analyzed (Participants) | 14
nanogram*hour per milliliter (ng*hr/mL) | 32010 (21)

7. Primary Outcome: PF-07321332 Average Plasma Concentration Over the Dosing Interval (Cav) on Day 10
Description: This was determined by AUCtau/tau.
Time Frame: Day 10 (pre-dose, 0.5, 1, 1.5, 2, 4, 6, 8, and 12 hours)
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram per milliliter (ng/mL)
Arm/Group | PF-07321332 300 mg + Ritonavir 100 mg
Number analyzed (Participants) | 14
nanogram per milliliter (ng/mL) | 2668 (21)

8. Primary Outcome: PF-07321332 Accumulation Ratio for AUCtau (Rac) on Day 10
Description: Accumulation ratio for AUCtau following multiple dosing was calculated as AUCtau on Day 10 divided by AUC12 on Day 1.
Time Frame: Day 1 (pre-dose, 0.5, 1, 1.5, 2, 4, 6, 8, and 12 hours); Day 10 (pre-dose, 0.5, 1, 1.5, 2, 4, 6, 8, and 12 hours)
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ratio
Arm/Group | PF-07321332 300 mg + Ritonavir 100 mg
Number analyzed (Participants) | 14
ratio | 1.627 (21)

9. Primary Outcome: PF-07321332 Accumulation Ratio for Cmax (Rac, Cmax) on Day 10
Description: Observed accumulation ratio for Cmax was calculated as Cmax on Day 10 divided by Cmax on Day 1.
Time Frame: Day 1 (pre-dose, 0.5, 1, 1.5, 2, 4, 6, 8, and 12 hours); Day 10 (pre-dose, 0.5, 1, 1.5, 2, 4, 6, 8 and 12 hours)
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ratio
Arm/Group | PF-07321332 300 mg + Ritonavir 100 mg
Number analyzed (Participants) | 14
ratio | 1.461 (22)

10. Primary Outcome: PF-07321332 Peak-to-trough Ratio (PTR) on Day 10
Description: This was determined by Day 10 Cmax/Day 10 Ctrough.
Time Frame: Day 10 (pre-dose, 0.5, 1, 1.5, 2, 4, 6, 8, and 12 hours)
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ratio
Arm/Group | PF-07321332 300 mg + Ritonavir 100 mg
Number analyzed (Participants) | 14
ratio | 4.517 (32)

11. Primary Outcome: PF-07321332 Apparent Clearance (CL/F) on Day 10
Description: Apparent oral clearance. This was determined by Dose/AUCtau.
Time Frame: Day 10 (pre-dose, 0.5, 1, 1.5, 2, 4, 6, 8, and 12 hours)
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liter/hour (L/h)
Arm/Group | PF-07321332 300 mg + Ritonavir 100 mg
Number analyzed (Participants) | 14
Liter/hour (L/h) | 9.379 (21)

12. Primary Outcome: PF-07321332 Apparent Volume of Distribution (Vz/F) on Day 10
Description: Apparent oral volume of distribution.
Time Frame: Day 10 (pre-dose, 0.5, 1, 1.5, 2, 4, 6, 8, and 12 hours)
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liters (L)
Arm/Group | PF-07321332 300 mg + Ritonavir 100 mg
Number analyzed (Participants) | 14
Liters (L) | 91.01 (29)

13. Primary Outcome: PF-07321332 Terminal Elimination Half-life (t½) on Day 10
Description: Terminal half-life. This was determined by Loge(2)/kel, where kel is the terminal phase rate constant calculated by a linear regression of the log-linear concentration-time curve.
Time Frame: Day 10 (pre-dose, 0.5, 1, 1.5, 2, 4, 6, 8, 12, 24 and 48 hours)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Hours (hr)
Arm/Group | PF-07321332 300 mg + Ritonavir 100 mg
Number analyzed (Participants) | 14
Hours (hr) | 6.842 (1.2336)

14. Primary Outcome: PF-07321332 Area Under the Plasma Concentration-time Profile From Time Zero to the Time of the Last Quantifiable Concentration (AUClast) on Day 10
Description: Area under the plasma concentration-time profile from time 0 to the time of the last quantifiable concentration (Clast)
Time Frame: Day 10 (pre-dose, 0.5, 1, 1.5, 2, 4, 6, 8, 12, 24 and 48 hours)
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram*hour per milliliter (ng*hr/mL)
Arm/Group | PF-07321332 300 mg + Ritonavir 100 mg
Number analyzed (Participants) | 14
nanogram*hour per milliliter (ng*hr/mL) | 41460 (24)

15. Primary Outcome: PF-07321332 Trough Concentration (Ctrough) on Day 5
Description: Concentration at pre-dose on Day 5. Observed directly from data.
Time Frame: Day 5 (pre-dose)
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram per milliliter (ng/mL)
Arm/Group | PF-07321332 300 mg + Ritonavir 100 mg
Number analyzed (Participants) | 14
nanogram per milliliter (ng/mL) | 1389 (26)

16. Primary Outcome: PF-07321332 Trough Concentration (Ctrough) on Day 8
Description: Concentration at pre-dose on Day 8. Observed directly from data.
Time Frame: Day 8 (pre-dose)
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram per milliliter (ng/mL)
Arm/Group | PF-07321332 300 mg + Ritonavir 100 mg
Number analyzed (Participants) | 14
nanogram per milliliter (ng/mL) | 1481 (27)

17. Primary Outcome: PF-07321332 Trough Concentration (Ctrough) on Day 10 (Pre-dose)
Description: Concentration at pre-dose on Day 10. Observed directly from data.
Time Frame: Day 10 (pre-dose)
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram per milliliter (ng/mL)
Arm/Group | PF-07321332 300 mg + Ritonavir 100 mg
Number analyzed (Participants) | 14
nanogram per milliliter (ng/mL) | 1333 (32)

18. Primary Outcome: PF-07321332 Trough Concentration (Ctrough) on Day 10 (12 Hours After Last Dose)
Description: Concentration at 12 hour time on Day 10. Observed directly from data.
Time Frame: Day 10 (12 hours after last dose)
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram per milliliter (ng/mL)
Arm/Group | PF-07321332 300 mg + Ritonavir 100 mg
Number analyzed (Participants) | 14
nanogram per milliliter (ng/mL) | 997.4 (40)

19. Secondary Outcome: Number of Participants With Treatment-Emergent Adverse Events (TEAEs)
Description: An adverse event (AE) is any untoward medical occurrence in a patient or clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. A serious AE was any untoward medical occurrence at any dose that resulted in death; was life-threatening; required hospitalization or prolongation of existing hospitalization; resulted in persistent or significant disability/incapacity; resulted in congenital anomaly/birth, was a suspected transmission via a Pfizer product of an infectious agent,pathogenic or non-pathogenic. An adverse event is considered a Treatment-Emergent Adverse Event (TEAE) if the event started during the effective duration of treatment. All events that started on or after the first dosing day and time/start time, if collected, but before the end of the study would be flagged as TEAEs.
Time Frame: From baseline up to Day 42
Population: The analysis population included all participants who took at least 1 dose of study intervention.
Measure: Count of Participants; unit: Participants
Arm/Group | PF-07321332 300 mg + Ritonavir 100 mg
Number analyzed (Participants) | 14
Participants
  TEAEs | 6
  serious TEAEs | 0

20. Secondary Outcome: Number of Participants With Vital Signs Data Meeting Pre-Specified Categorization Criteria
Description: Vital signs evaluations included supine blood pressure (BP) and pulse rate. The pre specified criteria for vital signs included systolic blood pressure (BP) minimum (min.) less than (<) 90 millimeter of mercury (mmHg); systolic BP change from baseline maximum (max.) decrease >= 30 mmHg, max. increase >=30 mmHg; diastolic BP min. <50mmHg; diastolic BP change from baseline max. decrease >=20, max. increase >=20; seated pulse rate min. <40 beats per minute (bpm) and max. >120 bpm. Participants who met at least 1 pre- specified criteria would be reported in outcome measure.
Time Frame: Day 1 (pre-dose, within 1-2 hours after morning dose), Day 10 (pre-dose, within 1-2 hours after morning dose)
Population: The analysis population included all participants who took at least 1 dose of study intervention.
Measure: Count of Participants; unit: Participants
Arm/Group | PF-07321332 300 mg + Ritonavir 100 mg
Number analyzed (Participants) | 14
Participants | 0

21. Secondary Outcome: Number of Participants With Laboratory Abnormalities
Description: Safety laboratory assessments included hematology, urinalysis, and clinical chemistry.
Time Frame: Day-1, Day 2, Day 5, Day 8, Day 10, Day 12.
Population: The analysis population included all participants who took at least 1 dose of study intervention.
Measure: Count of Participants; unit: Participants
Arm/Group | PF-07321332 300 mg + Ritonavir 100 mg
Number analyzed (Participants) | 14
Participants
  Urate (milligrams per decilitre[mg/dL]) > 1.2x upper limit of normal (ULN) | 2
  Fibrinogen (mg/dL) < 0.75x Baseline | 1
  Fibrinogen (mg/dL) > 1.25x Baseline | 2
  Urine Hemoglobin ≥ 1 | 2

22. Secondary Outcome: Number of Participants With Electrocardiogram (ECG) Data Meeting Pre-Specified Categorization Criteria
Description: The average of the triplicate readings collected at each assessment time was calculated for each ECG parameter. Baseline was defined as the average of the triplicate pre-dose recordings on Day 1. Pre-defined categories for corrected QT (Fridericia method) (QTcF): Absolute value (milliseconds[msec]) >450 and ≤480, or >480 and ≤500, or >500; Increase from baseline in QTcF (msec) >30 and ≤60, or>60. Pre-defined categories for PR and QRS: PR (msec) max. ≥300; PR (msec) increase from baseline: baseline >200 and max. ≥25% increase, or baseline ≤200 and max. ≥50% increase; QRS (msec) max. ≥140; QRS (msec) increase from baseline ≥50% increase. Participants who met at least 1 pre- specified criteria would be reported in outcome measure.
Time Frame: Day 1 (pre-dose, within 1-2 hours after morning dose), Day 10 (pre-dose, within 1-2 hours after morning dose)
Population: The analysis population included all participants who took at least 1 dose of study intervention.
Measure: Count of Participants; unit: Participants
Arm/Group | PF-07321332 300 mg + Ritonavir 100 mg
Number analyzed (Participants) | 14
Participants | 0

23. Secondary Outcome: Ritonavir Maximum Observed Plasma Concentration (Cmax) on Day 1
Description: Cmax is maximum plasma concentration
Time Frame: Day 1 (pre-dose, 0.5, 1, 1.5, 2, 4, 6, 8, and 12 hours)
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram per milliliter (ng/mL)
Arm/Group | PF-07321332 300 mg + Ritonavir 100 mg
Number analyzed (Participants) | 14
nanogram per milliliter (ng/mL) | 545.8 (50)

24. Secondary Outcome: Ritonavir Maximum Observed Plasma Concentration (Cmax) on Day 10
Description: Cmax is maximum plasma concentration
Time Frame: Day 10 (pre-dose, 0.5, 1, 1.5, 2, 4, 6, 8 and 12 hours)
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram per milliliter (ng/mL)
Arm/Group | PF-07321332 300 mg + Ritonavir 100 mg
Number analyzed (Participants) | 14
nanogram per milliliter (ng/mL) | 1109 (33)

25. Secondary Outcome: Ritonavir Time for Maximum Observed Plasma Concentration (Tmax) on Day 1
Description: Tmax is the time for maximum plasma concentration
Time Frame: Day 1 (pre-dose, 0.5, 1, 1.5, 2, 4, 6, 8 and 12 hours)
Population: as for outcome 1
Measure: Median (Full Range); unit: hours (hr)
Arm/Group | PF-07321332 300 mg + Ritonavir 100 mg
Number analyzed (Participants) | 14
hours (hr) | 2.00 [1.00 to 4.00]

26. Secondary Outcome: Ritonavir Time for Maximum Observed Plasma Concentration (Tmax) on Day 10
Description: Tmax is the time for maximum plasma concentration
Time Frame: Day 10 (pre-dose, 0.5, 1, 1.5, 2, 4, 6, 8 and 12 hours)
Population: as for outcome 1
Measure: Median (Full Range); unit: hours (hr)
Arm/Group | PF-07321332 300 mg + Ritonavir 100 mg
Number analyzed (Participants) | 14
hours (hr) | 2.00 [1.50 to 4.00]

27. Secondary Outcome: Ritonavir Area Under the Plasma Concentration-time Profile From Time Zero to Time Point on 12 Hours (AUC12) on Day 1
Description: This was determined by linear/Log trapezoidal method - reported as AUC12 on Day 1.
Time Frame: Day 1 (pre-dose, 0.5, 1, 1.5, 2, 4, 6, 8, and 12 hours)
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram*hour per milliliter (ng*hr/mL)
Arm/Group | PF-07321332 300 mg + Ritonavir 100 mg
Number analyzed (Participants) | 14
nanogram*hour per milliliter (ng*hr/mL) | 3136 (49)

28. Secondary Outcome: Ritonavir Area Under the Plasma Concentration-time Profile From Time Zero to Time Tau (Where Tau=12 Hours [Twice Daily Dosing]) (AUCtau) on Day 10
Description: as for outcome 6
Time Frame: Day 10 (pre-dose, 0.5, 1, 1.5, 2, 4, 6, 8, and 12 hours)
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram*hour per milliliter (ng*hr/mL)
Arm/Group | PF-07321332 300 mg + Ritonavir 100 mg
Number analyzed (Participants) | 14
nanogram*hour per milliliter (ng*hr/mL) | 6152 (29)

29. Secondary Outcome: Ritonavir Area Under the Plasma Concentration-time Profile From Time Zero to the Time of the Last Quantifiable Concentration (AUClast) on Day 10
Description: Area under the plasma concentration-time profile from time 0 to the time of the last quantifiable concentration (Clast)
Time Frame: Day 10 (pre-dose, 0.5, 1, 1.5, 2, 4, 6, 8, 12, 24, and 48 hours)
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram*hour per milliliter (ng*hr/mL)
Arm/Group | PF-07321332 300 mg + Ritonavir 100 mg
Number analyzed (Participants) | 14
nanogram*hour per milliliter (ng*hr/mL) | 7118 (33)

30. Secondary Outcome: Ritonavir Average Plasma Concentration Over the Dosing Interval (Cav) on Day 10
Description: This was determined by AUCtau/tau.
Time Frame: Day 10 (pre-dose, 0.5, 1, 1.5, 2, 4, 6, 8, and 12 hours)
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram per milliliter (ng/mL)
Arm/Group | PF-07321332 300 mg + Ritonavir 100 mg
Number analyzed (Participants) | 14
nanogram per milliliter (ng/mL) | 512.9 (29)

31. Secondary Outcome: Ritonavir Apparent Clearance (CL/F) on Day 10
Description: Apparent oral clearance. This was determined by Dose/AUCtau.
Time Frame: Day 10 (pre-dose, 0.5, 1, 1.5, 2, 4, 6, 8, and 12 hours)
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liter/hour (L/h)
Arm/Group | PF-07321332 300 mg + Ritonavir 100 mg
Number analyzed (Participants) | 14
Liter/hour (L/h) | 16.25 (29)

32. Secondary Outcome: Ritonavir Apparent Volume of Distribution (Vz/F) on Day 10
Description: Apparent oral volume of distribution. This was determined by Dose/(AUCtau*kel)
Time Frame: Day 10 (pre-dose, 0.5, 1, 1.5, 2, 4, 6, 8, and 12 hours)
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liters (L)
Arm/Group | PF-07321332 300 mg + Ritonavir 100 mg
Number analyzed (Participants) | 14
Liters (L) | 123.0 (23)

33. Secondary Outcome: Ritonavir Terminal Elimination Half-life (t½) on Day 10
Description: as for outcome 13
Time Frame: Day 10 (pre-dose, 0.5, 1, 1.5, 2, 4, 6, 8, 12, 24, and 48 hours)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Hours (hr)
Arm/Group | PF-07321332 300 mg + Ritonavir 100 mg
Number analyzed (Participants) | 14
Hours (hr) | 5.471 (1.7871)

34. Secondary Outcome: Ritonavir Trough Concentration (Ctrough) on Day 5
Description: Concentration at pre-dose on Day 5. Observed directly from data.
Time Frame: Day 5 (pre-dose)
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram per milliliter (ng/mL)
Arm/Group | PF-07321332 300 mg + Ritonavir 100 mg
Number analyzed (Participants) | 14
nanogram per milliliter (ng/mL) | 233.3 (38)

35. Secondary Outcome: Ritonavir Trough Concentration (Ctrough) on Day 8
Description: Concentration at pre-dose on Day 8. Observed directly from data.
Time Frame: Day 8 (pre-dose)
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram per milliliter (ng/mL)
Arm/Group | PF-07321332 300 mg + Ritonavir 100 mg
Number analyzed (Participants) | 14
nanogram per milliliter (ng/mL) | 212.8 (44)

36. Secondary Outcome: Ritonavir Trough Concentration (Ctrough) on Day 10 (Pre-dose)
Description: Concentration at pre-dose on Day 10. Observed directly from data.
Time Frame: Day 10 (pre-dose)
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram per milliliter (ng/mL)
Arm/Group | PF-07321332 300 mg + Ritonavir 100 mg
Number analyzed (Participants) | 14
nanogram per milliliter (ng/mL) | 200.8 (35)

37. Secondary Outcome: Ritonavir Trough Concentration (Ctrough) on Day 10 (12 Hours After Last Dose)
Description: Concentration at 12 hour on Day 10. Observed directly from data.
Time Frame: Day 10 (12 hours after last dose)
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram per milliliter (ng/mL)
Arm/Group | PF-07321332 300 mg + Ritonavir 100 mg
Number analyzed (Participants) | 14
nanogram per milliliter (ng/mL) | 134.9 (44)

ADVERSE EVENTS:
Time Frame: From baseline up to Day 42.
Description: The adverse events were reported by the treatment group of PF-07321332 300 mg + Ritonavir 100 mg, instead of by 2 treatment groups separately as PF-07321332 and ritonavir were dosed simultaneously (within no more than 5 minutes of each other).
Arm/Group | PF-07321332 300 mg + Ritonavir 100 mg
All-Cause Mortality (participants affected / at risk) | 0/14
Serious Adverse Events (participants affected / at risk) | 0/14
Other Adverse Events (participants affected / at risk) | 6/14
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | PF-07321332 300 mg + Ritonavir 100 mg (N=14)
Diarrhoea (Gastrointestinal disorders) | 4
Blood creatinine increased (Investigations) | 1
Rash (Skin and subcutaneous tissue disorders) | 1
Dysgeusia (Nervous system disorders) | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (2):
  • Study Protocol (2021-09-27): https://cdn.clinicaltrials.gov/large-docs/34/NCT05339334/Prot_000.pdf
  • Statistical Analysis Plan (2021-11-16): https://cdn.clinicaltrials.gov/large-docs/34/NCT05339334/SAP_001.pdf